CLINICAL TRIAL: NCT01631708
Title: Mi-Iron - Moderately Increased Iron - is Reducing Iron Overload Necessary?
Acronym: Mi-iron
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Austin Health (Other Government); Royal Brisbane and Women's Hospital (Other Government); Fremantle Hospital and Health Service (Other); Melbourne Health (Other); The University of Queensland (Other)
Responsible Party: Principal Investigator, Martin Delatycki, Professor, Murdoch Childrens Research Institute
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 04609
Record Dates: First submitted 2012-06-24; First posted 2012-06-29 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Hereditary Haemochromatosis
Keywords: Hereditary haemochromatosis; Moderate iron overload; Serum ferritin; Treatment
MeSH Terms: conditions — Hemochromatosis | interventions — Plasmapheresis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythrocytapheresis (Active Comparator): Erythrocytapheresis is a procedure whereby whole blood is drawn from an individual and all elements except erythrocytes are returned to the donor. An automated filtration process removes the erythrocytes.
  Those in arm 1 will have third weekly erythrocytapheresis until their SF is returned to the normal range.
  Interventions: Procedure: Erythrocytapheresis
- Plasmapheresis (Sham Comparator): In plasmapheresis, the plasma is removed by the automated filtration process whilst other blood elements including erythrocytes are returned to the subject.
  Those in arm 2 will have plasmapheresis with the approximate number of episodes of apheresis that would be required to reduce their SF to normal had they been randomised to the true treatment arm.
  Interventions: Procedure: Plasmapheresis

INTERVENTIONS:
Procedure: Erythrocytapheresis — To achieve a blinded randomised trial, apheresis treatment will be used. Those in arm 1 will have erythrocytapheresis reducing iron levels and those in arm 2 will have plasmapheresis and their iron levels will not be reduced.
  An apheresis machine will be used to remove red blood cells only from the erythrocytapheresis group. Subjects will have third weekly treatments until SF levels are reduced to ~100 ug/L in accordance with current guidelines.
  Other Names: red blood cell removal, red blood cell apheresis
  Arms: Erythrocytapheresis
Procedure: Plasmapheresis — An apheresis machine will be used to remove blood plasma only from the plasmapheresis group. Those in arm 2 will have the approximate number of episodes of apheresis that would be required to reduce their SF to normal had they been randomised to the true treatment arm. Those in the sham arm will be offered to have venesection at their choice of venue or to have their SF normalised by erythrocytapheresis after the initial blinded part of the study. This will be done because it will not be known for some time if there is benefit from normalisation of SF and therefore leaving people with elevated SF that may be harmful.
  Other Names: plasma removal, sham erythrocytapheresis
  Arms: Plasmapheresis

SUMMARY:
Haemochromatosis is a preventable genetic iron overload disorder. Untreated, it can shorten life due mainly to liver cirrhosis and cancer. It can be prevented by blood donation to maintain normal iron levels. It is unclear, however, whether treatment is necessary when individuals have moderate elevation of iron in the body. This research project will study the effects of treatment in this group by assessing a number of scans, questionnaires and blood tests in treated and untreated individuals.

DETAILED DESCRIPTION:
There is mounting evidence that treatment of moderate iron overload in HFE related hereditary haemochromatosis (HH) is not necessary. This project aims to undertake a randomised patient-blinded trial of erythrocytapheresis compared to sham erythrocytapheresis (using plasmapheresis) in individuals who have serum ferritin (SF) above the upper limit of the normal range but < 1000ug/L (defined here as moderate iron overload) due to HFE mutations and to compare the prevalence of symptoms and objective markers of disease in the two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. HFE C282Y homozygous.
2. Aged 18 - 70 years .
3. SF above the upper limit of the normal range of 300µg/L but less than 1000µg/L with a currently or previously raised TS (>greater than the upper limit of normal for the testing laboratory).

Exclusion Criteria:

1. HH due to genotypes other than HFE C282Y homozygosity.
2. Normal SF, SF > 1000µg/L.
3. Other major risk factor(s) for liver toxicity or other significant co-morbidities including positivity for hepatitis B or C, excess alcohol consumption (> 60g/day in males and 40g/day in females) or body mass index > 35.
4. Has had venesection therapy for HH in the last two years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Fatigue | Clinically and statistically significant change in measures taken at baseline and at the end of treatment will be compared. Patients will have approximately 6 third weekly treatments however this will vary depending on initial SF.
  Modified Fatigue Impact Scale (MFIS). The MFIS is a shortened version of the Fatigue Impact Scale. This 21-item scale can be self completed and measures the impact of fatigue on physical, cognitive and psychosocial functioning. Each item is scored from 0 (never) to 4 (almost always) resulting in a score from 0-84. In addition, physical (0-36), cognitive (0-40) and psychosocial (0-8) subscale scores can be derived.

SECONDARY OUTCOMES:
Change in markers of liver fibrosis | Clinically and statistically significant change in measures taken at baseline and at the end of treatment will be compared. Patients will have on average 6 third weekly treatments (15 weeks).
  Liver fibrosis will be assessed using Hepascore and Fibrometer (blood tests) and transient elastography (ultrasound).
Quality of life | Clinically and statistically significant change in measures taken at baseline and at the end of treatment will be compared. Patients will have on average 6 third weekly treatments (15 weeks).
  Medical Outcomes Study 36-item short form (SF36). As there are no specific quality of life tools available for HH, we will use this very widely used generic tool that has been used in a number of HH studies. This tool covers eight dimensions of health and wellbeing. One study found that individuals seen in a HH clinic and who had no clinical symptoms had significantly lower scores on a number of dimensions of the SF36 compared to population norms.
Depression and Anxiety | Clinically and statistically significant change in measures taken at baseline and at the end of treatment will be compared. Patients will have on average 6 third weekly treatments (15 weeks).
  The Hospital Anxiety and Depression Scale (HADS) is a brief self-report measure designed to screen for anxiety symptoms and depression symptoms in a hospital setting. It is composed of two seven-item subscales, the Anxiety (HADS-A) and Depression (HADS-D) subscales, and a 14-item total scale (HADS-T). Participants use a four-point Likert-type scale to rate how they have felt in the past week. It has been found to be valid and reliable in various populations.
Arthritis | Clinically and statistically significant change in measures taken at baseline and at the end of treatment will be compared. Patients will have on average 6 third weekly treatments (15 weeks).
  The presence and impact of arthritis will be measured by the Arthritis Impact Measurement Scales 2 short form. This is a 24 item validated scale that assesses the impact of arthritis on the individual over the past four weeks. We will also ascertain the use of arthritis medication at baseline and end of erythrocytapheresis/sham erythrocytapheresis.
Markers of oxidative stress | Clinically and statistically significant change in measures taken at baseline and at the end of treatment will be compared. Patients will have on average 6 third weekly treatments (15 weeks).
  To assess oxidative stress, we will measure F2-isoprostanes, a validated marker of cellular lipid oxidative damage, in urine and blood.

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Delatycki, Principal Investigator — Austin Health/Murdoch Childrens Research Institute
Locations (3):
- Australia (3):
  - Royal Brisbane and Woman's Hospital, Brisbane, Queensland
  - Austin Health, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria

REFERENCES:
- [Derived] Ong SY, Gurrin LC, Dolling L, Dixon J, Nicoll AJ, Wolthuizen M, Wood EM, Anderson GJ, Ramm GA, Allen KJ, Olynyk JK, Crawford D, Ramm LE, Gow P, Durrant S, Powell LW, Delatycki MB. Reduction of body iron in HFE-related haemochromatosis and moderate iron overload (Mi-Iron): a multicentre, participant-blinded, randomised controlled trial. Lancet Haematol. 2017 Dec;4(12):e607-e614. doi: 10.1016/S2352-3026(17)30214-4. PMID 29195602
- [Derived] Ong SY, Dolling L, Dixon JL, Nicoll AJ, Gurrin LC, Wolthuizen M, Wood EM, Anderson GJ, Ramm GA, Allen KJ, Olynyk JK, Crawford D, Kava J, Ramm LE, Gow P, Durrant S, Powell LW, Delatycki MB. Should HFE p.C282Y homozygotes with moderately elevated serum ferritin be treated? A randomised controlled trial comparing iron reduction with sham treatment (Mi-iron). BMJ Open. 2015 Aug 12;5(8):e008938. doi: 10.1136/bmjopen-2015-008938. PMID 26270952
- See also: Haemochromatosis Australia homepage — http://www.haemochromatosis.org.au/